CLINICAL TRIAL: NCT04282811
Title: An Observational Study to Evaluate the Clinical and Biologic Features and Outcome of Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) Treated With Venetoclax-based Regimens Outside Clinical Trials in Italy
Brief Title: Observational Study Relapsed or Refractory Chronic Lymphocytic Leukemia Venetoclax-based Regimens Outside Clinical Trials in Italy
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CLL1920
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Relapse Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort group: Patients who have received at least one dose of venetoclax
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Patients treated with venetoclax-based regimens outside clinical trials in Italy

SUMMARY:
Observational study aimed at describing the characteristics and outcome of CLL patients who started treatment with venetoclax-based regimens according to the local label outside clinical trials in Italy in a period of time ranging from the start of the Venetoclax Named Patient Program (March 2016) until June 30th, 2025.

DETAILED DESCRIPTION:
Observational study to describe the characteristics and outcome of CLL patients treated with venetoclax according to the local label. The study includes two different groups: a retrospective group (all patients who have received at least one dose of venetoclax before enrolment) and a prospective group (patients receiving treatment with venetoclax after enrolment). All patients in both groups will be observed for up to 48 months from the treatment start. In the prospective cohort only, QoL and treatment adherence will be assessed at the time of study entry (i.e. baseline) and thereafter at 3, 6, 9, 12, 18 24, 30, 36, 42 and 48 months of follow-up and at treatment discontinuation (due to any cause).

ELIGIBILITY:
Inclusion Criteria

1. Patients with R/R CLL fulfilling the eligibility criteria required by the Venetoclax Named Patient Program who have received at least 1 dose of venetoclax.
2. Patients with CLL who have received at least 1 dose of venetoclax or are scheduled to start treatment with venetoclax according to the Post-marketing Use before June 30th, 2025.
3. Signed informed consent document (if feasible) according to ICH/EU/GCP and national local laws indicating that the patients understand the purpose of the study and they agree to give complete access to their medical records.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients who started treatment with venetoclax-based regimens according to the local label outside clinical trials in Italy in a period of time ranging from the start of the Venetoclax Named Patient Program (March 2016) until June 30th, 2025.
Sampling Method: Probability Sample
Enrollment: 321 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of the PFS in relapsed/refractory (R/R) patients with CLL treated with venetoclax-based regimens according to the local label outside clinical trials in Italy. | 15 months
  Estimation of the PFS at 15 months from the start of venetoclax treatment in patients with R/R CLL who started treatment with venetoclax-based regimens according to the local label from the start of the Venetoclax Named Patient Program (March 2016) until October 31st, 2021

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona, Ferrara
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Ao Di Catanzaro "Pugliese-Ciaccio", Presidio Ospedaliero "Ciaccio - de Lellis" - Ematologia, Catanzaro
  - Ao Di Cosenza, Presidio Ospedaliero Annunziata - Uoc Ematologia, Cosenza
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Irccs Ospedale S. Raffaele - Milano - Unità Neoplasie Linfocitarie B, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Ausl Della Romagna, Ospedale "Santa Maria Delle Croci" - Ravenna - Ematologia, Ravenna
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" Po E. Morelli - Reggio Calabria - Uoc Ematologia, Reggio Calabria
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Ao S. Maria - Terni - Sc Onco Ematologia, Terni
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Asst Dei Sette Laghi, Ospedale Di Circolo E Fondazione Macchi - Uoc Ematologia, Varese
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona